CLINICAL TRIAL: NCT04321551
Title: Clinical Trial of Androgen Effects on the Reproductive Neuroendocrine Axis
Brief Title: Hormone Secretion in Transgender Males
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study not funded in previous iteration. new clinicaltrials.gov protocol submitted for funded version of study
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tracy Harrison, Professor of Obstetrics, Gynecology, and Reproductive Sciences, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200395
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Transgender; Healthy
Keywords: Testosterone therapy
MeSH Terms: interventions — testosterone 17 beta-cypionate; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Provocative Hormonal Testing (Experimental): TGN subjects will undergo baseline endocrine and menstrual cycle evaluation, followed by intramuscular (i.m.) administration of testosterone cypionate (TC) 50 mg (standard dose) every 7 d for 32 wks (Fig. 8). After 24 wks, an aromatase inhibitor, letrozole (LET, 2.5 mg/d oral), will be co-administered with TC for 8 wks to block estrogen synthesis and examine whether T's effects are independent of E2 signaling.
  Interventions: Drug: Testosterone Cyp 200Mg/Ml Inj (in Oil); Drug: Letrozole

INTERVENTIONS:
Drug: Testosterone Cyp 200Mg/Ml Inj (in Oil) — Depo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)- cyclopentylpropionate ester of the androgenic hormone testosterone. Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1- oxopropoxy)-, (17ß)-. Its molecular formula is C27H40O3, and the molecular weight 412.61.
  Other Names: Depo-Testosterone
Drug: Letrozole — Letrozole is a nonsteroidal aromatase inhibitor (inhibitor of estrogen synthesis). It is chemically described as 4,4'-(1H-1,2,4-Triazol-1- ylmethylene)dibenzonitrile. Letrozole is a white to yellowish crystalline powder, practically odorless, freely soluble in dichloromethane, slightly soluble in ethanol, and practically insoluble in water. It has a molecular weight of 285.31, empirical formula C17H11N5, and a melting range of 184°C to 185°C. Letrozole is available as 2.5 mg tablets for oral administration.
  Other Names: Femara

SUMMARY:
Aim 1 utilizes prospective clinical studies in TGN to test the hypothesis that prolonged exogenous androgens alter menstrual cyclicity by inhibiting gonadotropin secretion, steroid hormone release, and ovulation. We will utilize a clinical trial of TRT to evaluate T suppression of ovarian follicle and hormone dynamics (Aim 1A) and LH pulsatility (Aim 1B).

DETAILED DESCRIPTION:
We will conduct a prospective, controlled clinical trial of ovarian and menstrual cyclicity in TGN initiating TRT (Fig. 8). Enrollment will include 30 TGN and 30 cisgender female (CF) control subjects who report female gender identity congruent with female sex assignment at birth. All subjects will be age >18 y, with female sex assignment at birth, regular menstrual cycles, and body mass index 18-35 kg/m2. Subjects with history of prior T use, cancer, chemotherapy, or radiation of the brain, abdomen, or pelvis, current use of hormonal medications (including, but not limited to, metformin, insulin, progestins, or estrogenic medications), current endocrinopathy (including, but not limited to, PCOS, androgen secreting tumor, diabetes, or pituitary, thyroid, or adrenal disease), and renal, hepatic, cardiac, or hematologic disease will be excluded. TGN subjects will undergo baseline endocrine and menstrual cycle evaluation, followed by intramuscular (i.m.) administration of testosterone cypionate (TC) 50 mg (standard dose) every 7 d for 32 wks (Fig. 8). After 24 wks, an aromatase inhibitor, letrozole (LET, 2.5 mg/d oral), will be co-administered with TC for 8 wks to block estrogen synthesis and examine whether T's effects are independent of E2 signaling. TGN will collect first morning-voided urine daily at home for assessment of hormone levels during one complete menstrual cycle before TRT begins and continuing during TRT during wks 8-12, 20-24 and 28-32 . Untreated CF controls will collect urine daily during one menstrual cycle. Urinary concentrations of LH, FSH, estrone (E1) conjugates, and pregnanediol glucuronide (PdG) will be measured via ELISA. Studies of steroidogenesis during the menopausal transition have demonstrated accuracy of monitoring urinary hormone metabolite levels to reconstruct ovarian cyclicity and ovulatory patterns; we can use this methodology to track progression of any declining HPG axis output over time. All subjects will complete a daily uterine bleeding log using REDCap® and undergo weekly measurement of serum FSH, LH, E2, and P4 (ELISA), and T (LC-MS/MS) for confirmation of hormone dynamics demonstrated by urine hormone metabolite studies. TGN will also undergo weekly transvaginal ultrasound (US) using a 4- to 9-MHz probe to obtain three-dimensional (3D) pelvic imaging following initiation of TRT for confirmation of corpus luteum (CL) formation and regression analysis of hormone secretion patterns, endometrial thickness, antral follicle count (AFC), and volume of the uterus and ovaries. Changes in follicle dynamics will be studied with 3D US determination of the mean diameter of each antral in 1-mm increments from 2 to 9 mm, as in our prior reports.

The primary endpoint will be Evidence of Luteal Activity (ELA), as defined by a 3-fold increase in urinary PdG level over baseline. Basal urinary PdG levels, normalized to urinary creatinine excretion, will be determined based upon the minimum daily PdG level detected per cycle or 4-wk interval, as previously described. Secondary endpoints will include mean serum FSH and LH levels, peak urinary LH concentration, and cumulative LH surge count. Follicular phase function will be defined per cycle (or per 4-wk interval in amenorrheic subjects) by creatinine-adjusted urinary E1 AUC. Five-day moving averages of creatinine-adjusted urinary FSH and LH levels will be calculated, with LH surge defined as a 3 standard deviation increase in the 5-d moving LH average, as previously described. The proportion of subjects demonstrating an LH surge will be compared during successive 4-wk intervals.

We have already demonstrated successful recruitment and retention of TGN and CF participants in longitudinal studies involving daily urine collection and serial pelvic US (e.g., our study in Fig. 2 and others). TGN subjects will be serially evaluated for adverse effects of TRT per The Endocrine Society recommendations. Details regarding safety monitoring are in the Human Subjects Section.We calculate that 20 subjects/group will have >95% power to detect a 30% decrease in the proportion of subjects with ELA at baseline compared to the final 4-wk TC study interval (wks 21-24). Although we anticipate a larger, more clinically meaningful decrease, we utilized a conservative target to maximize the study's power. While we have had no dropouts in our current TGN pilot study, a 1/3 dropout rate is factored into our enrollment target of 30 subjects/group to ensure achieving sufficient power. Although we anticipate a larger, more clinically meaningful decrease, we have utilized a conservative target to maximize the study's power.

ELIGIBILITY:
* Self-identified transgender or non-binary person assigned female at birth
* No history of prior testosterone therapy
* Regular menstrual cycles
* Body mass index 18 - 35
* Hemoglobin greater than than 11 gm/dl at screening evaluation
* Presence of uterus and both ovaries at time of consent
* Able to provide informed consent
* No current endocrine disease- including, but not limited to, pituitary disease, adrenal disease, androgen secreting tumor, polycystic ovary syndrome, diabetes, or untreated thyroid disease.
* Absence of cancer and any renal, hepatic, or cardiac disease
* No current use of endocrine modulating medications (including, but not limited to, progestin therapy, estrogen containing medications, metformin, insulin)
* No history of radiation or surgery involving brain, abdomen, or pelvis

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender females Transgender males Gender non-binary individuals
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evidence of Luteal Activity | Baseline, 12 weeks, 24 weeks, and 32 weeks
  The primary endpoint will be Evidence of Luteal Activity (ELA), as defined by a 3-fold increase in urinary pregnanediol glucuronide level over baseline.

IPD SHARING:
Plan to Share IPD: No